CLINICAL TRIAL: NCT07353086
Title: Evaluation of Horizontal Mandibular Ridge Augmentation Through Subperiosteal Tunneling by Using Bovine Sticky Bone (Radio-Histological Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Rasha Yousif Mohamed Elsayed, Principal investigator, Tanta University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-4-24-2180.
Record Dates: First submitted 2026-01-13; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Posterior Mandible With Deficient Ridge Width
Keywords: ridge augmentation ,subperiosteal tunneling , sticky bone

STUDY DESIGN:
Intervention Model Description: Single group assignment Participants in this study received horizontal mandibular ridge augmentation using an enriched bovine bone graft matrix (sticky bone) through the subperiosteal tunneling technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Horizontal Mandibular Ridge Augmentation through Subperiosteal Tunneling by Using Bovine sticky bone (Experimental): Participants underwent ridge augmentation with enriched bovine sticky bone delivered through subperiosteal tunneling in the posterior mandible
  Interventions: Procedure: Ridge augmentation with enriched bovine sticky bone through the subperiosteal tunneling technique in the posterior mandible

INTERVENTIONS:
Procedure: Ridge augmentation with enriched bovine sticky bone through the subperiosteal tunneling technique in the posterior mandible — Under local anesthesia, a 5-mm vertical incision was made in the attached gingiva remote from the augmentation site. A primary subperiosteal tunnel was then created using a microsurgical periosteal elevator and further extended with VISTA tunneling elevators from the Mitex VISTA Tunneling Kit (No. 1-6) for less accessible areas. Multiple cortical perforations were subsequently performed using a Piezo surgery® UI1 tip (1.6 mm) to enhance vascularity. Bovine sticky bone was delivered via a modified insulin syringe for precise placement, condensed using a bone condenser, and excess material was removed from the incision site. The graft was molded upward against the cortical bone to eliminate dead spaces. CGF membranes were placed over the graft site to support healing, followed by closure with simple interrupted sutures

SUMMARY:
This clinical trial evaluated horizontal ridge augmentation in the posterior mandible using subperiosteal tunneling with enriched bovine bone graft matrix (sticky bone). The minimally invasive procedure addressed horizontal bone deficiencies without flap elevation, while preserving periosteal integrity and reducing patient morbidity. Ten patients underwent clinical assessment of wound healing, pain, and neurosensory changes over 4 weeks; radiological evaluation of CBCT-measured bone width at immediate postoperative and 6-month follow-up; and histological analysis of bone core biopsies obtained at implant placement to evaluate remodeling and graft integration.

DETAILED DESCRIPTION:
The alveolar bone is a tooth-dependent tissue that extends from the basal bone of the maxilla and mandible to form and support the tooth sockets. Resorption of alveolar bone may be attributed to a variety of factors, such as tooth loss, trauma, periodontal disease, and pathologies. Tooth loss is often followed by a bone remodeling process leading to gradual horizontal and vertical bone ridge reduction.

The posterior mandible is the most challenging region for reconstruction and implant placement due to its critical neurovascular structures, thick cortical bone, and reduced vascular trabecular bone, requiring careful treatment planning for successful outcomes Multiple techniques such as osteoplasty, narrow implants, bone augmentation, ridge splitting, and distraction osteogenesis address deficient ridge width. However, conventional augmentation in the posterior mandible requires flap elevation and barrier membranes, increasing risks of complications such as pain, swelling, wound dehiscence, and membrane exposure.

To address these limitations, this study employed the subperiosteal tunneling technique for horizontal augmentation of posterior edentulous ridges. By creating a subperiosteal pouch without extensive flap elevation, this approach reduces tissue trauma, preserves periosteal integrity essential for bone regeneration, and eliminates the need for barrier membranes by harnessing the periosteum's regenerative potential.

Bovine sticky bone was utilized for its cohesive properties, enhanced stability, and regenerative potential. (31) This study evaluated the radiological and histological outcomes of horizontal mandibular ridge augmentation through subperiosteal tunneling using enriched bovine bone graft matrix (sticky bone). Conducted at the outpatient clinic of the Oral and Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University.

Ten adult patients with mandibular horizontal alveolar ridge atrophy were included in the study. Their ages ranged from 34 to 42 years (mean ± SD: 38 ± 2.6). The gender distribution was 40% male and 60% female participants, reflecting women's predominance in dental treatment-seeking behavior.

At the 6-month follow-up, subperiosteal tunneling with sticky bone achieved a 90% success rate (9/10 patients). One 41-year-old female patient experienced failure (10%) due to an intraoperative tear during crestal tunneling, resulting in soft tissue compromise, infection, dehiscence, and total graft loss. The remaining patients demonstrated successful bone formation, rapid soft tissue healing with minimal morbidity, no dehiscence or graft exposure, and excellent long-term outcomes, confirming this technique's reliability as a membrane-free ridge augmentation alternative.

Clinical assessment of postoperative healing, using the Landry et al. healing index (161), demonstrated predictable progression from predominantly good healing at one week (60%) to universal excellent healing by one month, maintained through six months, which indicates a transient inflammatory response and a favorable biocompatibility and healing profile for the procedure.

Pain levels, assessed by the Visual Analog Scale (VAS), declined substantially throughout the treatment period. The mean VAS score was 3.70 ± 1.42 at one week, which significantly decreased to 1.30 ± 0.82 at two weeks. From the third week onward no pain was reported, with mean VAS scores consistently at 0 ± 0. Neurosensory function remained preserved throughout the follow-up period in all patients.

Radiographic assessment at six months demonstrated significant horizontal ridge augmentation with a mean width gain of 3.30 ± 0.97 mm. The calculated resorption rate of 17.58 ± 4.76% remained within biologically acceptable parameters for horizontal ridge augmentation procedures.

Histological examination of bone core specimens obtained during implant placement revealed Hematoxylin and Eosin (H&E)-stained sections showing graft remnants well-integrated with mature lamellar bone, without evidence of inflammation or necrosis. Woven bone exhibited plump osteoblasts indicative of active bone formation, sparse osteoclasts with minimal resorption, and multiple reversal lines confirming ongoing remodeling. Osteoconduction was evident with graft particles surrounded by osteogenic cells and newly formed bone. Immunohistochemical analysis demonstrated strong osteocalcin expression within the bone matrix and moderate cytoplasmic staining in osteocytes of newly formed bone, confirming active mineralization and robust bone remodeling activity.

ELIGIBILITY:
Inclusion Criteria:

1. Adequate vertical ridge height but less than 4 mm of bone width in the posterior mandible, which required bone grafting.
2. Patients who were motivated, cooperative, and had good oral hygiene.

Exclusion Criteria:

1. Any uncontrolled systemic disease or medications that might compromise. healing, osseointegration or complicate the surgical procedures such as uncontrolled diabetes.
2. Presence of fenestrations or dehiscence of the residual wall.
3. Smoking habit of 20 cigarettes or more per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-08-25 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Horizontal Bone Gain in mm | 6 months postoperatively
  The horizontal bone gain was measured radiographically using CBCT imaging to evaluate the effectiveness of ridge augmentation with enriched bovine sticky bone through subperiosteal tunneling in the posterior mandible."

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Shoushan, Professor of OMFS, Study Director — Faculty of Dentistry ,Tanta university ,Egypt; Dalia H Zahran, Professor of oral Biology, Principal Investigator — Faculty of Dentistry ,Tanta university ,Egypt; Maram N Breshah, Lecturer of OMFS, Principal Investigator — Faculty of Dentistry ,Tanta university ,Egypt
Locations (1):
- Faculty of Dentisty ,university of Tanta, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared to protect participant privacy and confidentiality. The small sample size in this surgical study increases re-identification risk

REFERENCES:
- Available data/document: Informed Consent Form: rasha-yousif@hotmail.com — https://dent.tanta.edu.eg/post-forms.aspx